CLINICAL TRIAL: NCT06428643
Title: A Seek, Test, and Treat Intervention to Reduce Chlamydia Trachomatis Disparities in Black Youth Living in the Deep South
Brief Title: A Seek, Test, and Treat Intervention to Reduce Chlamydia Trachomatis Disparities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Patricia Kissinger, Principal Investigator, Tulane University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-377
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Chlamydia; Gonorrhea; Hiv; Syphilis
Keywords: Screening; Expedited Treatment
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Acquired Immunodeficiency Syndrome; Syphilis | interventions — HIV Testing

STUDY DESIGN:
Intervention Model Description: Community based screening of young men for chlamydia, gonorrhea, HIV, and syphilis. Expedited treatment for positive subjects and their sexual partners.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chlamydia, gonorrhea, syphilis, and HIV screening (Experimental): Community screening of individuals for chlamydia and gonorrhea is not normally done. We are testing to see if this intervention will impact the rates of chlamydia among women.
  Interventions: Other: Chlamydia, gonorrhea, syphilis, and HIV screening

INTERVENTIONS:
Other: Chlamydia, gonorrhea, syphilis, and HIV screening — Individuals aged 15-26 years old will be tested for chlamydia, gonorrhea, HIV, and syphilis at community based venues. Individuals who test positive for chlamydia and gonorrhea and their sexual partners will be offered expedited treatment at participating pharmacies. Individuals who test positive will be asked to be rescreened for Ct/GC at 3 months post treatment.

SUMMARY:
This study includes testing for four STIs (chlamydia, gonorrhea, syphilis, and HIV) at no cost. If positive, individual subjects will also be counseled and offered options for treatment for themselves and their sex partners that may include no cost expedited treatment and the option to be rescreened 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as African American or Black
* 15-26 years of age
* Lives or spends most of their time in Orleans Parish
* Had vaginal sex at least once

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Unable to speak or understand English
* Previously enrolled in the study
* Known to be pregnant
* Known HIV positive status

Ages: 15 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2322 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of chlamydia in women | up to 60 months
  Primary outcome

SECONDARY OUTCOMES:
Rate of gonorrhea in women | up to 60 months
  Secondary outcome

IPD SHARING:
Plan to Share IPD: No